CLINICAL TRIAL: NCT07019714
Title: Clinical Research on the Improvement of Exercise Endurance in Idiopathic Pulmonary Fibrosis by Daoyin Technique
Brief Title: Daoyin Technique for Improving Exercise Endurance in IPF
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Liaoning University of Traditional Chinese Medicine (Other)
Collaborators: The First Affiliated Hospital of Henan University of Traditional Chinese Medicine (Other); Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Daoyin for IPF
Record Dates: First submitted 2025-06-05; First posted 2025-06-13 (Actual); Last update posted 2025-06-13 (Actual); Status verified 2025-05

CONDITIONS: Idiopathic Pulmonary Fibrosis
Keywords: Idiopathic Pulmonary Fibrosis; Daoyin Technique; randomized controlled trial
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daoyin Technique in addition to the guideline - directed treatment. (Experimental): The experimental group was given Daoyin Technique in addition to the treatment guided by the guideline "Idiopathic Pulmonary Fibrosis (an Update) and Progressive Pulmonary Fibrosis in Adults: An Official ATS/ERS/JRS/ALAT Clinical Practice Guideline "
  Interventions: Behavioral: Daoyin Technique
- Routine Comprehensive Training in addition to the guideline - directed treatment. (Active Comparator): The experimental group was given routine Comprehensive Training in addition to the treatment guided by the guideline "Idiopathic Pulmonary Fibrosis (an Update) and Progressive Pulmonary Fibrosis in Adults: An Official ATS/ERS/JRS/ALAT Clinical Practice Guideline "
  Interventions: Behavioral: Routine Comprehensive Training

INTERVENTIONS:
Behavioral: Daoyin Technique — On the basis of treatment guided by "Idiopathic Pulmonary Fibrosis (an Update) and Progressive Pulmonary Fibrosis in Adults: An Official ATS/ERS/JRS/ALAT Clinical Practice Guideline ", the experimental group was given Daoyin Technique for treatment. For patients who are able to complete the respiratory guidance technique. For patients who are unable to complete the respiratory guidance technique but have stable vital signs (referring to the "Expert Consensus on Respiratory Critical Care Rehabilitation Treatment Techniques in China"), the supine guidance technique is selected. It is carried out 5 days a week, 2 times a day, and each training session lasts for 30 minutes.
  Arms: Daoyin Technique in addition to the guideline - directed treatment.
Behavioral: Routine Comprehensive Training — On the basis of treatment guided by I"Idiopathic Pulmonary Fibrosis (an Update) and Progressive Pulmonary Fibrosis in Adults: An Official ATS/ERS/JRS/ALAT Clinical Practice Guideline",the experimental group was given Routine Comprehensive Training. According to the patient's condition, select aerobic training (such as walking) or upper - limb and lower - limb resistance training (such as lifting, chest - expanding, foot - pedaling movements, etc.) combined with respiratory training (such as pursed - lip breathing, abdominal breathing, etc.). The heart rate should reach the target heart rate range and last for more than 10 minutes. This training is carried out 5 days a week, 2 times a day.
  Arms: Routine Comprehensive Training in addition to the guideline - directed treatment.

SUMMARY:
This study is based on the previously constructed digital rehabilitation management platform, scientifically evaluating the clinical efficacy of guided technology in improving IPF exercise endurance, and forming high-quality clinical evidence.

DETAILED DESCRIPTION:
This study is based on a digital and intelligent rehabilitation management platform. It collects patients' movement data through intelligent motion capture equipment and heart rate, blood oxygen, and other data using fitness trackers, to complete rehabilitation tracking management, real-time assessment, and effect evaluation. Adopting a multi-center,non inferiority, randomized controlled clinical trial design, 236 IPF patients were selected as the research subjects. Based on the guideline-directed treatment, the experimental group received guided techniques, while the control group received conventional comprehensive training. The intervention lasted for 3 months, followed by a 3-month follow-up. The primary outcome measures were 6MWD and 30- second sit-to-stand test, while secondary outcome measures included acute exacerbation, FVC, DLCO, VO2 peak, mMRC score, ATAQ-IPF score, etc. The study elucidated the mechanism of action, scientifically evaluated the impact of guided techniques on IPF endurance, and established a guided technique protocol for IPF.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who meet the diagnostic criteria for IPF;
2. Those who can tolerate guided - technique training;
3. Aged between 40 and 85 years old;
4. Those who can independently or with the assistance of family members use devices such as smartphones and computers during home - based training;
5. Those who voluntarily accept treatment and sign the informed consent form.

Exclusion Criteria:

1. Patients in the acute exacerbation phase of IPF.
2. Patients with comorbidities such as chronic obstructive pulmonary disease, lung cancer, active pulmonary tuberculosis, bronchiectasis, pulmonary embolism, and other pulmonary diseases.
3. Patients with severe cardiovascular and cerebrovascular diseases (malignant arrhythmia, unstable angina pectoris, acute myocardial infarction, cardiac function at grade 3 or above, stroke, cerebral hemorrhage, etc.).
4. Patients with severe liver diseases (such as bleeding caused by liver cirrhosis, portal hypertension, and esophagogastric varices) and severe kidney diseases (dialysis, kidney transplantation, etc.).
5. Patients with severe osteoarthropathy or osteoporosis, and those with unstable fractures.
6. Patients with progressive neuromuscular diseases.
7. Patients with unclear consciousness, dementia, and various mental illnesses.
8. Pregnant or lactating women, and patients with a recent pregnancy plan.
9. Patients who have been participating in other clinical trials within 1 month before enrollment.
10. Patients who need long - term use of ventilators and those with unstable vital signs while bedridden.

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 236 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2028-06-30 (Estimated); Study Completion 2028-12-30 (Estimated)

PRIMARY OUTCOMES:
6 Six Minute Walk Distance(6MWD) | Change from baseline 6MWD at week 13 and 26.
  6MWD will be applied to evaluate the exercise capacity. The higher values indicate the better exercise capacity.
the 30 - second sit - to - stand test(30s STS) | Change from baseline FVC at week 13 and 26.
  30s STS will be used to assess pulmonary function.

SECONDARY OUTCOMES:
The time of the first acute exacerbation | Up to week 26.
  The time of the patients' first acute exacerbation will be recorded.
Frequency of acute exacerbation | Up to week 26.
  Frequency of acute exacerbation will be recorded.
Frequency of acute exacerbations resulting in hospitalization | Up to week 26.
  Frequency of acute exacerbation resulting in hospitalization will be recorded.
Frequency of acute exacerbations resulting in ICU admission | Up to week 26.
  Frequency of acute exacerbation resulting in ICU admission will be recorded.
Forced vital capacity (FVC) | Change from baseline FVC at week 13 and 26.
  FVC will be used to assess pulmonary function.
Forced expiratory volume in one second(FEV1) | Change from baseline FEV1 at week 13 and 26.
  FEV1 will be used to assess pulmonary function.
Percent of FEV1#FEV1%# | Change from baseline FEV1% at week 13 and 26.
  FEV1% will be used to assess pulmonary function.
Diffusing Capacity of Carbon Monoxide#DLCO# | Change from baseline DLCO at week 13 and 26.
  DLCO will be used to assess pulmonary function.
Cardiopulmonary Exercise Testing(CPET) | Change from baseline Peak Oxygen Uptake, Anaerobic Threshold, Breathing Reserve, and ventilatory equivalent for carbon dioxide at week 13 and 26.
  CPET will be used to evaluate the cardiopulmonary function of the human body during exercise. Parameters such as Peak Oxygen Uptake, Anaerobic Threshold, Breathing Reserve, and ventilatory equivalent for carbon dioxide will be collected.
Blood oxygen saturation(SpO2) | Change from baseline SpO2 at week 13 and 26.
  SpO2 of the subjects is measured by a finger clip pulse oximeter.
Dyspnea | Change from baseline mMRC scores at week 13 and 26.
  Dyspnea will be assessed by 22.modified Medical Research Council(mMRC) scores. A score of 0-4 will be given according to the degree of immediate dyspnea. A higher score indicates a worse condition.
A Tool to Assess Quality of life (ATAQ-IPF) | Change from baseline ATAQ-IPF scores at week 13 and 26.
  ATAQ - IPF is currently a specialized scale for evaluating the quality of life of patients, consisting of 13 dimensions and 74 items, with each item being scored from 1 to 5 points. A higher score indicates a worse condition.
St. George's respiratory questionnaire (SGRQ) | Change from baseline SGRQ scores at week 13 and 26.
  SGRQ is a scale used to evaluate the quality of life of patients, which includes three dimensions: symptoms, mobility, and the impact of disease on daily life, with a total of 50 items. A higher score indicates a worse condition.
Clinical symptoms and Signs | Change from baseline clinical symptoms and signs up at week 13 and 26.
  Clinical symptoms and Signs will be evaluated through a scale. The scale includes coughing, expectoration, chest tightness, shortness of breath, wheezin. The Clinical Symptom Rating Scale includes 6 items: cough, expectoration, chest tightness, shortness of breath, wheezing, and cyanosis. Each item has a score of 0-3, totaling 18 points. The higher the score, the worse he patient's condition.
Imaging findings | Up to week 13, 26.
  Imaging findings will bedetected by High - Resolution Computed Tomography (HRCT) of the chest.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Liaoning University of Traditional Chinese Medicinenese Medicine, Shenyang, Liaoning, China